CLINICAL TRIAL: NCT02453633
Title: Theory Based SMS Reminders - Text's Impact on Patient Attendance
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Lovisenberg Diakonale Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: SMS-ENT
Record Dates: First submitted 2015-05-21; First posted 2015-05-25 (Estimated); Last update posted 2015-05-25 (Estimated); Status verified 2015-05

CONDITIONS: Otorhinolaryngologic Diseases; Sleep Disorders; Hearing Disorders
Keywords: Appointment reminder; Attendance; No-show
MeSH Terms: conditions — Otorhinolaryngologic Diseases; Sleep Wake Disorders; Hearing Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Emotional SMS text (Experimental): Patients in this arm will receive an emotion-based SMS reminder of their scheduled outpatient clinic appointment.
  Interventions: Other: Emotional SMS text
- Standard SMS text (Active Comparator): Patients in this arm will receive the standard SMS reminder of their scheduled outpatient clinic appointment.
  Interventions: Other: Standard SMS text

INTERVENTIONS:
Other: Emotional SMS text — SMS appointment reminder with the following text (translated from Norwegian):
  Reminder about your appointment. There are many who are waiting for treatment. Please notify us if you can not make your appointment on: Tuesday 31 March at 10:00.
  tel. 23225501 or send email to kirpolonh@lds.no later than one weekday prior to your appointment.
  No-show fee: Kr. 640.
  Lovisenberg Diakonale Hospital, Department of Surgery, Ear, Nose and Throat. Do not reply to this message per SMS.
  Arms: Emotional SMS text
Other: Standard SMS text — SMS appointment reminder with the following text (translated from Norwegian):
  Reminder of appointment at Lovisenberg Diakonale Hospital, Department of Surgery, Ear, Nose and Throat: Wednesday 11.feb 2015 at 10:00. For a change, call tel. 23225501 or send email to kirpolonh@lds.no. Do not reply to this message per SMS.
  Arms: Standard SMS text

SUMMARY:
The project will be done at the ear, nose and throat outpatient department at Lovisenberg Diakonale Hospital (LDS) in 2015-2016. About 12% of patients with appointments at the surgical outpatient clinic at LDS do not attend their appointment even after receiving both letters and shot message service (SMS) reminders. Persuasion theory suggests that the SMS reminders may be more effective if the text appeals more to the patient's feelings. The project is designed as a randomized controlled trial in which the control group receives the standard text that has neutral content and the intervention group receives a more emotion-based SMS reminder. The aim is to determine whether the more emotional text reduces the proportion of patients who do not show up for their scheduled appointment at the surgical outpatient clinic.

DETAILED DESCRIPTION:
Studies from Norway's Health South East (HSØ) show that the number of patients who do not attend their scheduled appointments account for 200 000 to 250 000 outpatient consultations each year. For comparison, there are 270,000 patients waiting for treatment. It has thus been recommended that regional health authorities take measures to reduce the number of patients who do not attend their scheduled appointment.

This study will evaluate whether short message service (SMS) appointment reminders that appeal to the patient's emotions are more effective for reducing non-attendance to scheduled outpatient appointments at the ear, nose, and throat outpatient clinic at Lovisenberg Diakonale Hospital in Oslo, Norway. The study will be designed as randomized controlled trial in which 2000 patients are randomly assigned to either the intervention group (emotional SMS text) or the control group (standard SMS text with neutral content). Because theory suggests that emotion-based text messages will be more effective reminders, it is hypothesized that they will result in a 50% reduction in the number of patients who do not show for their appointment compared to the control group.

ELIGIBILITY:
Inclusion Criteria:

* Patients (any diagnosis) with a scheduled clinic appointment at the LDS Ear, Nose and Throat Surgical Clinic or scheduled for polysomnography during the inclusion period.
* Date of birth on or after 01.01.1935

Exclusion Criteria:

* Patients with 2 appointments on the same day, only the first appointment will be included.
* Patients without a phone number
* Patients born before 01.01.1935
* Included patients will not be included again if they get a new appointment in the inclusion period.

Max Age: 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2000 (Estimated)
Dates: Start 2015-05; Primary Completion 2015-08 (Estimated); Study Completion 2015-08 (Estimated)

PRIMARY OUTCOMES:
Appointment attendance | Day of scheduled appointment
  Patient attendance at their scheduled clinic appointment (yes = show up at or before the scheduled time or reschedule at least 24 hours before appointment; no=does not show up by the appointed time).

CONTACTS AND LOCATIONS:
Overall Officials: Bjørn Holm, MD, Study Director — Lovisenberg Diakonale Hospital; Anners Lerdal, RN, PhD, Principal Investigator — Lovisenberg Diakonale Hospital